CLINICAL TRIAL: NCT04280484
Title: Evaluating the Use of Acute Intermittent Hypoxia to Improve Symptoms in Persons With Multiple Sclerosis
Brief Title: Acute Intermittent Hypoxia in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Milap Sandhu, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU00207024
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Intermittent Hypoxia (Experimental): 1 minute of 9% oxygen in the inspired air, alternating with 1 minute of 21% oxygen; for a total of 15 bouts
  Interventions: Other: Intermittent Hypoxia
- Sham Acute Intermittent Hypoxia (Sham Comparator): 1 minute of 21% oxygen in the inspired air, alternating with 1 minute of 21% oxygen; for a total of 15 bouts.
  Interventions: Other: Sham Hypoxia

INTERVENTIONS:
Other: Intermittent Hypoxia — 1 minute of 9% oxygen in the inspired air, alternating with 1 minute of 21% oxygen; for a total of 15 iterations/episodes.
  Arms: Acute Intermittent Hypoxia
Other: Sham Hypoxia — 1 minute of 21% oxygen in the inspired air, alternating with 1 minute of 21% oxygen; for a total of 15 iterations/episodes.
  Arms: Sham Acute Intermittent Hypoxia

SUMMARY:
The overall objective of this project is to investigate the effectiveness of Acute Intermittent Hypoxia (AIH), to improve muscle strength and activity level in individuals with relapsing-remitting MS.

ELIGIBILITY:
Inclusion Criteria:

* Have relapsing-remitting MS
* Volitional ankle plantar flexion strength in at least one leg
* Are relapse free for 30 days
* Patient-Determined Disease Steps scale score between 3 and 5 (3=gait disability to 5=late cane, need cane to walk 25 feet)

Exclusion Criteria:

* Currently taking antispasticity medications,
* Have cardiovascular or respiratory/pulmonary disorders, metabolic dysfunction, or prior diagnoses of obstructive sleep apnea
* Pregnant or nursing women (safety for developing fetus or infant is unknown)
* Cognitive concerns (must be able to consent to study, follow steps)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Voluntary Ankle Strength | 60 minutes post-intervention
  Maximum isometric ankle plantar-flexion and dorsi-flexion torque using a Biodex

SECONDARY OUTCOMES:
Electromyogram activity | 60 minutes post-intervention
  Plantar-flexor and Dorsi-flexor electromyogram activity
Symbol Digit Modalities Test | 60 minutes post-intervention
  The symbol-digit modalities test (SDMT) is a symbol substitution neuropsychological test that examines a person's attention and speed of processing

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States